CLINICAL TRIAL: NCT05300412
Title: The Role of Interleukin-7 Serum Level as Biological Marker in Breast Cancer: a Cross-sectional, Observational, and Analytical Study
Brief Title: The Role of Interleukin-7 Serum Level as Biological Marker in Breast Cancer
Status: Completed | Type: Observational
Sponsor: University Clinical Centre of Kosova (Other)
Responsible Party: Principal Investigator, Faton sermaxhaj, Medical Doctor, University Clinical Centre of Kosova
Other Study IDs: grid.412416.4
Record Dates: First submitted 2022-03-18; First posted 2022-03-29 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Breast Cancer Invasive
Keywords: Breast cancer, interleukins, interleukin-7, biomarker
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study has been to explore whether there is any elevation of Interleukin-7 serum level in the early invasive breast cancer (EIBC) patients in comparison with healthy controls. In addition the correlation between the Interleukin-7 serum level and histopathological characteristics of the tumor, has been evaluated.

We have hypothesized that Interleukin-7 serum level is elevated in the patients diagnosed with early invasive BC in comparison with healthy control group, and positively correlates with the tumor size, poor cell differentiation, lymphovascular and perineural invasion, negative hormone receptors' status, axillary lymph node metastasis, and the high Ki-67 proliferation index. In addition, no difference in the Interleukin-7 serum level exists between the patients recruited in Croatia and Kosovo, respectively.

This cross-sectional, observational, and analytical study has included 213 consecutive patients with EIBC (113 from Croatia and 100 from Kosovo) and 62 healthy participants as the control group (30 from Croatia and 32 from Kosovo). Blood samples have been taken from patients confirmed with breast cancer (BC) by biopsy, prior to surgical intervention and other oncological treatments, as well as from healthy participants. Interleukin-7 serum level has been measured, using "Sandwich" ELISA Immunoenzyme test. In addition, after the surgical intervention, the histopathological specimen examinations and the immunohistochemistry have been performed and analyzed. The differences of the distribution of the numerical variables have been analyzed with Mann-Whitney U test and Kruskal-Wallis ANOVA test. Correlations have been tested with Pearson coefficients. P value <0.05 has been accepted as statistically significant.

DETAILED DESCRIPTION:
This cross-sectional, observational, and analytical study has been undertaken in the Clinic of Oncology, University Hospital Center Zagreb, Croatia, and the Department of Thoracic Surgery in the University Clinical Center of Kosovo in Prishtina, Kosovo, from June 2018 until December 2019. In order to determine the Interleukin-7 serum level, blood samples (10 ml venous blood) have been taken from 213 EIBC patients, from which 100 from Kosovo University Hospital and 113 from Croatian University Hospital, prior to surgery and other oncological treatments, such as chemotherapy, radiotherapy, endocrine therapy or target therapy. On the other hand, the blood samples (10 ml venous blood) have been taken also from other 62 healthy participants, which compose the control group, from whom 32 from Kosovo and the other 30 from Croatia. Blood samples categorized in tubes have been identifiable only by the numbers attributed to participants, and have been stored frozen in temperatures of -20˚C, in order to conduct the analysis later.

Patients have been selected as consecutive among women, aged between 20 - 70 who are confirmed to BC, by biopsy, operable and without distant metastases. Patients with pathological conditions, such as acute and/or chronic inflammatory diseases, rheumatoid disease and other malignancies occurring simultaneously, patients receiving immune modulatory therapy, patients previously treated by surgery, chemotherapy, radiotherapy, target therapy or endocrine therapy, patients with dementia or any other psychological disorders unable to willingly participate in the study, have been excluded. The control group has been composed by women, aged between 20 - 70, without breast tumors, confirmed by ultrasound or mammography in the last three months or any other confirmed malignancies, without any acute or chronic inflammatory disease as well as no receiving immune modulatory therapy.

In this study, the Interleukin-7 serum level has been measured, using "Sandwich" ELISA Immunoenzyme test, human Interleukin-7 antibody, and Platinum ELISA using research tools from eBioscience Inc., located in San Diego, CA USA. After the surgery (partial or modified radical mastectomy) with or without axillary lymph node dissection or sentinel lymph node biopsy (SLNB), the histopathological specimen examinations have been performed according to routine practice, and the histopathological and immunohistochemistry features have been evaluated. Cancer staging has been conducted according to tumor node metastasis (TNM)-classification, by the American Joint Committee on Cancer Classification (AJCC). The patients have been classified in accordance to their pathological characteristics, including tumor size, histological types, histological grade, LVI and PNI, metastatic lymph nodes, molecular markers such as; ER, PR, amplification of Her-2/neu, Ki-67 proliferation index, molecular surrogate subtypes according to the St Gallen consensus criteria. The data on age and menopausal status have been also obtained from the patients.

Interleukin-7 serum level has been initially determined in all the study participants, including patients and the control group. Then it has been evaluated if there has been any difference of Interleukin-7 serum level between EIBC patients and control group. After that, appropriate analyzes have been done to see if there is any correlation between Interleukin-7 serum level of the patients and histopathological characteristics of the tumor, as well as age and menopausal status. In addition, the potential difference of Interleukin-7 serum level between patients coming from Croatia and Kosovo has been evaluated.

After checking for normality of distribution, numerical variables have been presented as median and interquartile range. The differences of the distribution of the numerical variables have been analyzed with Mann-Whitney U test and Kruskal-Wallis ANOVA test. Associations between numerical variables have been analyzed as Spearman rank correlation coefficient. Analyses have been performed with statistical software SPSS-22.0. The diagnostic accuracy and the optimal cut point value for Interleukin-7 level between two groups have been obtained based on the value of the area under the ROC curve.

ELIGIBILITY:
Inclusion Criteria:

* Patients with invasive breast cancer, confirmed with biopsy
* Operable and without distant metastases.

Exclusion Criteria:

* Patients with acute and/or chronic inflammatory diseases, rheumatoid disease and other malignancies occurring simultaneously
* Patients receiving immune modulatory therapy
* Patients previously treated by surgery, chemotherapy, radiotherapy, target therapy or endocrine therapy
* Patients with dementia or any other psychological disorders unable to willingly participate in the study.

Exclusion Criteria for the control group:

* Breast tumors or any other confirmed malignancies
* Any acute or chronic inflammatory disease
* Receiving immune modulatory therapy

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In order to determine the Interleukin-7 serum level, blood samples (10 ml venous blood) have been taken from 213 EIBC patients, from which 100 from Kosovo University Hospital and 113 from Croatian University Hospital, prior to surgery and other oncological treatments, such as chemotherapy, radiotherapy, endocrine therapy or target therapy. On the other hand, the blood samples (10 ml venous blood) have been taken also from other 62 healthy participants, which compose the control group, from whom 32 from Kosovo and the other 30 from Croatia. Blood samples categorized in tubes have been identifiable only by the numbers attributed to participants, and have been stored frozen in temperatures of -20˚C, in order to conduct the analysis later.
  Patients have been selected as consecutive among women, aged between 20 - 70. Also, the control group has been composed by women, aged between 20 - 70.
Sampling Method: Probability Sample
Enrollment: 275 (Actual)
Dates: Start 2018-06-05 (Actual); Primary Completion 2019-09-10 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Interleukin-7 | 7 days
  The amount of Interleukin-7 in the blood of the patients is determined in units (pg/ml), and is done using "Sandwich" ELISA Immunoenzyme test, human Interleukin-7 antibody, and Platinum ELISA using research tools from eBioscience Inc., located in San Diego, CA USA.

SECONDARY OUTCOMES:
Tumor size | 2 months
  The tumor size is determined by units (cm)
Histological type of tumor | 2 months
  The tumors are classified in these histological types: Invasive ductal carcinoma, invasive lobular carcinoma and others.
Histological grade | 2 months
  Based on histological grade the tumors are classified as: G1, G2, G3.
Lymphovascular and perineural invasion | 2 months
  Based on the lymphovascular and perineural invasion, the tumors are divided in positive or negative.
Metastatic lymph nodes | 2 months
  First, all the patients are divided in two groups: involved metastatic lymph nodes and without involved lymph nodes. After that, the involved cases are divided as: N1, N2, N3, based on the number of positive lymph nodes.
Molecular markers: Estrogen, progesterone, Her2/neu, Ki-67 proliferation index. | 2 months
  ER, PR, Her-2 status and Ki-67 proliferation index were interpreted according to the criteria of the American Society of Clinical Oncology (ASCO) and St. Gallen International Expert Consensus. According to these recommendations, ER and PR are considered positive if ≥1% of tumor cell nuclei exhibit a positive reaction. According to the same criteria, Her-2/neu expression by immunohistochemistry may range from 0 to 3. If the result is 0 to 1, it is considered negative. In contrast, if the result is 3, it is considered positive. Cases with a value of 2 are considered equivocal and are subject to fluorescent in situ hybridization (FISH) or chromogenic in situ hybridization (CISH) analysis. The Ki-67 value was determinated as percentage, from (1 - 100)%.
Molecular surrogate subtypes of Breast cancer | 2 months
  Based on the St. Gallen Consensus there are five molecular surrogate subtypes of invasive BC according to the expression of formerly mentioned molecular markers, namely, Luminal A-like, Luminal B/Her-2 negative-like, Luminal B/Her-2 positive-like, Her-2 positive type and Triple negative.
Age | 2 months
  The patients are divided based on the age
Menopausal status | 2 months
  Based on menopausal status patients are divided in premenopausal and postmenopausal.

CONTACTS AND LOCATIONS:
Overall Officials: Besim Sermaxhaj, MD, Principal Investigator — University Clinical Center Kosovo
Locations (1):
- Faton I. Sermaxhaj, MD, Pristina, Kosovo